CLINICAL TRIAL: NCT01054118
Title: Sitagliptin Combo Study
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Doses of JNJ-38431055, Sitagliptin, and Co-administration of JNJ-38431055 and Sitagliptin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR016348
Record Dates: First submitted 2010-01-15; First posted 2010-01-22 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 001 (Experimental): JNJ-38431055 Liquid suspension of JNJ-38431055 administered as a single dose
  Interventions: Drug: JNJ-38431055
- 002 (Active Comparator): Sitagliptin 100 mg Capsule containing 100 mg of sitagliptin administered as a single dose
  Interventions: Drug: Sitagliptin 100 mg
- 003 (Experimental): JNJ-38431055 + Sitagliptin 100 mg Liquid suspension of JNJ-38431055 administered as a single dose and capsule containing 100 mg of sitagliptin administered as a single dose
  Interventions: Drug: JNJ-38431055 + Sitagliptin 100 mg
- 004 (Placebo Comparator): Placebo Placebo suspension and placebo capsule administered as single doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-38431055 — Liquid suspension of JNJ-38431055 administered as a single dose
  Arms: 001
Drug: Sitagliptin 100 mg — Capsule containing 100 mg of sitagliptin administered as a single dose
  Arms: 002
Drug: JNJ-38431055 + Sitagliptin 100 mg — Liquid suspension of JNJ-38431055 administered as a single dose, and capsule containing 100 mg of sitagliptin administered as a single dose
  Arms: 003
Drug: Placebo — Placebo suspension and placebo capsule administered as single doses
  Arms: 004

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics (explores what the body does to the drug), and pharmacodynamics (explores what a drug does to the body) of single doses of JNJ-38431055, sitagliptin, and co-administration of JNJ-38431055 and sitagliptin in healthy overweight or obese adult male volunteers.

DETAILED DESCRIPTION:
This is a double-blind (neither physician or volunteer knows the name of the assigned study drug), placebo controlled (substance containing no medication), study in healthy, overweight or obese adult male volunteers. For each volunteer, the study consists of a screening phase (up to 30 days), a treatment phase during which volunteers will receive 4 study treatments in a randomized (study sequence assigned by chance) sequence (28 days), and a follow-up phase (10 days). During the treatment phase there will be at least 7 days between each of the 4 treatments. The four treatments will be JNJ-38431055, sitagliptin, JNJ-38431055 and sitagliptin, and placebo. The following safety evaluations will be taken throughout the study: Electrocardiogram (an ECG is a painless procedure that gives a picture of the electrical activity of the heart), blood pressure, heart rate, and blood samples for laboratory tests. The primary outcome will be the effect of JNJ-38431055 and sitagliptin on glucagon like peptide-1 (GLP-1) levels. Study drug will be administered as single oral doses separated by at least 7 days. The four treatments will be JNJ-38431055, sitagliptin, JNJ-38431055 and sitagliptin, and placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 27.0 and 38.0 kg/m2 (inclusive)
* Healthy on the basis of physical examination including medical history, vital signs, 12-lead ECG, and all other screening lab tests
* Men must agree to use a double barrier method of birth control (e.g., condom for them and use of spermicide with diaphragm, hormonal contraceptives or intrauterine devices by female partner) during the study and for three months following the last dose of study medication, and to not donate sperm during the study and for 3 months after receiving the last dose of study medication

Exclusion Criteria:

* History of, or currently active, illness or medical condition or disorder that the Investigator considers to be clinically significant
* Smoker or tobacco user within the past 6 months
* History of recent major surgery (within 6 months of study start)
* Positive test for alcohol and/or drugs of abuse
* Psychological and/or emotional problems, which would render the informed consent invalid, or limit the ability of the volunteer to comply with the study requirements
* Any condition that, in the opinion of the investigator, would compromise the well being of the volunteer or the study or prevent the volunteer from meeting or performing study requirements

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-12; Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
GLP-1 levels after a standard meal | 0-4 hours after the standard meal

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics of JNJ-38431055 administered alone and in combination with sitagliptin. | 24 hours after dosing
Assess the effect of JNJ-38431055 on appetite and satiety using a visual analogue scale (VAS) | Within 24 hours of dosing
Assess the safety and tolerability of JNJ-38431055 administered alone and in combination with sitagliptin as measured by occurrence of adverse events, ECGs, vital signs, and safety laboratory measurements. | From screening visit through follow-up visit
Assess incremental glucose changes after a meal tolerance test (MTT) | 0-4 hours after MTT

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (1):
- Lincoln, Nebraska, United States